CLINICAL TRIAL: NCT03674008
Title: A Phase III,Randomized, Double-blind, Propofol-controlled, Parallel-design, Multi-center Study Evaluating The Efficacy and Safety of HSK3486 for Sedation or Anesthesia in Patients Undergoing Colonoscopy and Gastroscopy
Brief Title: A Phase III Study Evaluating The Efficacy and Safety of HSK3486 for Sedation or Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK3486-301
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-07

CONDITIONS: Sedation or Anesthesia
Keywords: Sedation anesthesia gastrointestinal endoscopy
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): 0.4mg/kg/0.2 mg/kg
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): 1.5mg/kg/0.75mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — HSK3486 intravenous (iv) 0.4 mg/kg for induction, and 0.2 mg/kg top-ups for maintenance.
  Arms: HSK3486
Drug: Propofol — Propofol iv 1.5 mg/kg for induction, and 0.75 mg/kg top-ups for maintenance.
  Arms: Propofol

SUMMARY:
This is a Phase III, randomized, double-blind, propofol-controlled, parallel-design, multi-center study to evaluate the efficacy and safety of HSK3486 for sedation or anesthesia in patients undergoing colonoscopy and gastroscopy.

The study will enroll approximately 280 adults. The maximum study duration is anticipated to be up to nine months.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a diagnostic or therapeutic colonoscopy or gastroscopy;
2. Male or female patients, ASA grade I~II, aged ≥ 18 and < 65;
3. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2;
4. During screening and baseline, the respiratory rate ≥10 and ≤24, SpO2 when inhaling ≥95%, SBP≥90mmHg, DBP≥60mmHg, HR≥60 and ≤100;
5. Patient can understand the procedure of this study and is willing to comply with study requirements. The patient can sign the ICF voluntarily.

Exclusion Criteria:

1. Patients were contraindicated in general anesthesia.
2. Patients with a known sensitivity to propofol, opioids, naloxone, eggs, soy products or a medical condition such that these agents were contraindicated.
3. The patient has some history or evidence of increased risk of sedation or anesthesia, such as cardiovascular disease, respiratory disease, cerebrovascular disease, gastrodintestinal disease and other system disease prior to the screening and/or baseline period.
4. Patients with a history of drug or ethanol abuse with the past 3 months.
5. Patients with respiratory management difficulties (Modified Mallampati grade IV).
6. Patients in receipt of any investigational drug within 30 days before screening.
7. Patients in receipt of propofol, opioid , other sedative or anesthetic or analgesics within 72 hours prior to baseline.
8. Abnormal laboratory results consisting of any of the following:

1) neutrophil count≤ 1.5×109/L； 2）platelet≤ 80×109/L； 3）hemoglobin≤ 90 g/L; 4）aspartate aminotransferase≥ 1.5×ULN； 5）total bilirubin≥ 1.5×ULN； 6） serum creatinine≥ 1.2×ULN. 9. Pregnant women or female patients with a positive serum or urine human chorionic gonadotropin pregnancy test at screening or baseline or lactating female patients.

10. Patients with an inability to communicate well with the investigator, or deemed unsuitable according to the investigator (in each case providing a reason).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Success of colonoscopy procedure | from the first dose of the study drug to removal of colonoscope on day 1
  Measured by completion of colonoscopy, no requirement for an alternative sedative or anesthesia drug and no requirement for more than 5 doses of study drug within any 15 minute period.

SECONDARY OUTCOMES:
The success rate of the gastroscopy procedure | from the first dose of the study drug to removal of gastroscope on day 1
The success rate of the colonoscopy and gastroscopy procedure | from the first dose of the study drug to rem oval of colonoscope and gastroscope on day 1
Time to induction of sedation or anaesthesia | from the first dose of the study drug to the first MOAA/S scores≤1 on day 1
Time to start of procedure | From first dose of study drug until insertion of colonoscope or gastroscope on day 1
Time to fully alert | from the removal of colonoscopy or gastroscopy procedure, until the first of three consecutive MOAA/S scores of 5 on day 1
Time to discharge | from the removal of colonoscopy or gastroscopy procedure, until the first of three consecutive Aldrete scores of more than or equal to 9 on day 1
Sedation/anesthesia satisfaction, satisfaction assessment of subjects, anesthesiologists, and endoscopic physicians | from time to fully alert, until time to discharge on day 1

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Changde, China